CLINICAL TRIAL: NCT04503642
Title: Impact of Changing the Surgical Team for Wound Closure on Surgical Site Infection: a Matched Case-control Study
Brief Title: Changing the Surgical Team for Wound Closure and Surgical Site Infection
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: CLOT-T trial
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Incidence of Surgical Site Infection; Morality; Fascial Hernia
Keywords: Surgical Site Infection; Changing the surgical team
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: The intervention consisted in the closure of the abdominal wall and skin by a second surgical team which included a board-certified surgeon and a resident.
  Interventions: Procedure: Changing the surgical team for wound closure
- Baseline Group: During the baseline period, closure of the abdominal wall was performed by the main surgical team, the same team that performed the whole surgery.

INTERVENTIONS:
Procedure: Changing the surgical team for wound closure — The intervention consists of the exchange of the primary surgical team with a second surgical team that consists of one surgeon and one student. The first surgical team then may leave the operation theatre but is continuously accessible for questions.
  Groups: Intervention Group

SUMMARY:
Surgical site infection is a frequent complication after abdominal surgery. The wound closure is done at the end of the procedure when the attention of the entire team may be affected because of tiredness and reduced attention of the surgical team.

With this study, the investigators aim to test if an exchange of the surgical team by a specialised wound closure team may reduce the impact of surgical site infection.

ELIGIBILITY:
Inclusion Criteria:

* General Consent as documented by signature
* Patients undergoing elective or emergency abdominal surgery from Monday to Friday with wound closure from 8:00 until 17:30 and duration of operation.
* Age over 18 years

Exclusion Criteria:

* Patients < 18 years of age
* Patients with preexisting SSI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Visceral Surgery of the University Hospital Bern, a tertiary care centre
Sampling Method: Non-Probability Sample
Enrollment: 1160 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with SSIs | 30 days postoperative
  SSI that occur after surgery will be assessed according to the criteria developed by the Centers for Disease Control and Prevention. Infections will be categorized as incisional (superficial or deep) infections or organ-space infections. Superficial SSI (type 1) involve only skin and subcutaneous tissue and exclude stitch abscesses. Deep SSI (type 2) involve deeper soft tissues, like fascia and muscle, at the site of incision. Organ-space SSI (type 3) involve any organ or body cavity

SECONDARY OUTCOMES:
Postoperative Mortality at 30 days | 30 days postoperative
  Observer receives the information during the follow-up phone call that the patient died. If patients do not respond to follow-up phone calls, five documented attempts to contact the patients followed by rapid contacts with the subject's general practitioner or other medical staff involved in the medical treatment of the patients, will be performed before loss to follow-up is documented. In addition, the Zivilstandsamt will be contacted once 3 months after surgery.
Numbers of patients with fascial dehiscence at 30 days postoperative | 30 days postoperative
Numbers of patients with complications | 30 days postoperative
  Assessment according to Clavien-Dindo grading

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, MD, Principal Investigator — Visceral and transplant sugery, university hospital Berne
Locations (1):
- Dep. of Visceral and transplant surgery, Berne University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Salm L, Chapalley D, Perrodin SF, Tschan F, Candinas D, Beldi G. Impact of changing the surgical team for wound closure on surgical site infection: A matched case-control study. PLoS One. 2020 Nov 5;15(11):e0241712. doi: 10.1371/journal.pone.0241712. eCollection 2020. PMID 33151978